CLINICAL TRIAL: NCT01929915
Title: Perioperative Epidural Analgesia for Short-term and Long-term Outcomes of Pancreatic Cancer Surgery- Randomised Trial
Brief Title: Analgesia and Pancreatic Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201203094RIC
Record Dates: First submitted 2013-07-18; First posted 2013-08-28 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fentanyl; Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural patient controlled analgesia (Active Comparator): Epidural patient controlled analgesia
  Interventions: Procedure: Epidural patient controlled analgesia
- Intravenous patient controlled analgesia (Sham Comparator): Intravenous patient controlled analgesia for post operative pain control
  Interventions: Drug: Intravenous patient controlled analgesia

INTERVENTIONS:
Procedure: Epidural patient controlled analgesia — Patient controlled epidural analgesia with marcaine(1mg/ml)+ fentanyl(1.25mcg/ml)for postoperative pain control
  Other Names: Fentanyl; marcaine(bupivacaine hydrochloride)
  Arms: Epidural patient controlled analgesia
Drug: Intravenous patient controlled analgesia — Intravenous patient controlled analgesia with morphine(1mg/ml)for post operative pain control
  Other Names: morphine
  Arms: Intravenous patient controlled analgesia

SUMMARY:
Long-term survival for patients with pancreatic carcinoma is low, even following resection, the 5-year survival rate of patients ranges from 10 to 25%1. Most treatment failure is due to local recurrence, distant metastasis or both within one to two years after surgery2-4.

Surgery has been suggested to accelerate the development of preexisting micro metastases and to promote the establishment of new metastases5. Release of catecholamine and proinflammatory products secondary to surgical stress is believed to promote cancer progression6. Maintenance of proper anesthetic depth is beneficial to attenuate surgical stress. However, general anesthesia including numerous induction agents, volatile anesthetics and opioids, is associated with immunosuppression especially on the cell-mediated immunity which has a crucial role in prevention of micrometastasis5,7. Therefore, regional anesthesia and analgesia which effectively attenuating surgical stress while efficiently reducing general anesthetics consumption, seem to provide promising advantages to prevent perioperative cancer progression. Currently, most studies available in humans are retrospective and observational to evaluate regional anesthesia and prostate, colorectal, breast and cervical cancer-related outcomes8-12. Only one randomized study investigating major abdominal cancer surgery is available13. However, it is not specific to an individual cancer type and perioperative cell-mediated immunity is not evaluated.

In this study, we aimed to identify whether epidural block beneficial to early surgical and late cancer-related outcomes in patients receiving pancreatic cancer surgery. Perioperative cell-mediated immunity functions including natural killer cells, helper and cytotoxic T-lymphocytes were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer expected to receive curative Whipple operation

Exclusion Criteria:

* palliative operation
* preoperative chemotherapy or radiotherapy
* patients with metastasis
* contraindications for epidural catheter placement
* prior spine surgery

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Perioperative immunoprofile | one week
  Immunoprofile measurements: CD4+, CD8+, CD19+, NK cells, Dendritic cells, regularoty T cells

SECONDARY OUTCOMES:
survival rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Cheng Chan, M.D., Principal Investigator — Department of Anesthesiology, NTUH, Taipei, Taiwan
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Cummings KC 3rd, Xu F, Cummings LC, Cooper GS. A comparison of epidural analgesia and traditional pain management effects on survival and cancer recurrence after colectomy: a population-based study. Anesthesiology. 2012 Apr;116(4):797-806. doi: 10.1097/ALN.0b013e31824674f6. PMID 22273991